CLINICAL TRIAL: NCT05071196
Title: Impact of Facilitated Vegan Diet on Cardiometabolic Endpoints and Trimethylamine N-oxide
Brief Title: Facilitated Vegan Diet on Cardiometabolic Endpoints and Trimethylamine N-oxide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Pham, Principal Investigator, David Grant U.S. Air Force Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWH20210097H
Record Dates: First submitted 2021-09-02; First posted 2021-10-08 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cardiometabolic Risk Factors
Keywords: Vegan; boxed meal kit; trimethylamine N-oxide; cardiometabolic

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitated Vegan Diet (Experimental): The facilitated vegan participants will self-prepare and consume 2 vegan meal kits per day for 4 weeks
  Interventions: Other: Facilitated Vegan Diet
- Standard Omnivorous Diet (Active Comparator): The standard omnivorous arm will self-prepare and consume 2 non-vegan meal kits per day for 4 weeks
  Interventions: Other: Omnivorous Diet

INTERVENTIONS:
Other: Facilitated Vegan Diet — Vegan boxed meal kits
  Arms: Facilitated Vegan Diet
Other: Omnivorous Diet — Non-vegan boxed meal kits
  Arms: Standard Omnivorous Diet

SUMMARY:
Vegan meal kit delivery offers consumer convenience and has shown benefit in cardiometabolic parameters such as low-density lipoprotein cholesterol (LDL-c) and weight. The purpose of this study is to evaluate the impact of meal kit facilitated vegan diet on LDL-c and trimethylamine N-oxide (TMAO) when compared to an omnivorous diet control.

DETAILED DESCRIPTION:
This study will compare the impact of a vegan diet to a non-vegan diet, when provided with meal kits in participants who are overweight.

A vegan diet includes foods that come from plants and excludes foods that come from animals like meat, dairy, and eggs. Dietary modifications such as adopting a vegan diet are associated with significant improvements in cardiometabolic parameters, making it one of the preferred treatment options for obesity and preventing associated health conditions. Meal kits are packages that include: a quick (~30-45 minutes) and simple recipe, all the recipe's required ingredients, and are conveniently delivered to patient homes. In this study, a facilitated vegan diet is defined as a change from an omnivorous diet to a vegan diet with the aid of boxed vegan meal kit delivery. A facilitated vegan diet has shown LDL-c and weight improvements over continuing an omnivorous diet in a preliminary study.

TMAO, changes in gut microbiome, and compliance to dietary modification impact cardiovascular and overall health. TMAO is a diet dependent biomarker for CVD, as elevated TMAO levels are associated with a 62% increased risk of heart attack, stroke, or death. TMAO increases platelet hyperactivity, inflammation, and foam cell generation, all of which contribute to atherosclerosis and may explain the increased risk of CVD. Additionally, TMAO predicts risk of major adverse cardiovascular events independently of other cardiovascular risk factors.

Consumption of animal products elevate TMAO levels due to its abundance of TMAO precursors: choline and carnitine. Chronic dietary red meat was associated with increased TMAO levels over white meat and non-meat protein. One study found that consuming plant-based alternative meat products improved TMAO levels over a mostly red meat diet. Both study interventions replaced protein sources but did not remove animal products such as eggs and dairy, which have conflicting evidence relative to TMAO. This study intervention will have participants adopt a full vegan diet, eliminating animal products.

The gut microbiome plays a crucial role in converting dietary precursors into TMAO. TMAO levels post l-carnitine ingestion were significantly higher in patients on a long-term omnivorous diet vs patients on a long-term vegan or vegetarian diet. This suggests that the gut microbiome in a plant-based diet lowers the formation of TMAO via the diet. This study will explore changes in gut microbiome from a dietary intervention in relation to TMAO and explore if these changes are sustained after discontinuing a 4-week facilitated vegan diet. Additionally, changes in gut microbiome will be explored in relation to microbiota changes seen in other disease states such as anxiety, irritable bowel disease, and other inflammatory diseases.

The impact of dietary modifications on controlling obesity and associated health conditions has room for improvement. Dietary modifications have long been one of the preferred treatments in obesity and CVD prevention, yet the obesity rates continue to rise. One potential area of improvement is compliance to dietary modification. This study will explore changes in food group restricted free diet patterns after a 4-week vegan meal kit intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* BMI ≥ 25kg/m^2
* Consume ≥ 5 servings red meat per week
* Active duty military and Department of Defense (DoD) Beneficiaries with active Tricare insurance
* Willing and able to adopt a vegan or standard omnivorous diet for 4 weeks
* Willing and able to track meal patterns, nutritional intake, exercise activity, and adverse events for 13 weeks
* Willing and able to come to David Grant USAF Medical Center for 4 blood draws
* Able to receive weekly emails and receive and prepare meal kits

Exclusion Criteria:

* Currently on a vegetarian, vegan, or food-group restricted diet
* Currently taking or planning to initiate medications or supplements that significantly affect TMAO levels, carnitine, choline, or gut microbiome (Systemic antibiotics, antifungals, antivirals, antiparasitic, corticosteroids, methotrexate, cytokines, or immunosuppressive cytotoxic agents, laxatives, proton pump inhibitors, resveratrol, meldonium, or metformin)
* Currently consuming the following ≥ 2 times per week: probiotics/prebiotics, probiotic enhanced foods (eg. enhanced yogurt, kefir, kombucha), or energy drinks, multivitamins, or supplements with choline, carnitine, or betaine (Acceptable to consume: non-probiotic enhanced yogurts, energy drinks and multivitamins without choline, carnitine, or betaine)
* Participants will have the option to delay study start if they express interest in the study and have permanently discontinued one of the excluded diet, medication, or supplement listed previously within the past 4 weeks (minimum 4 week time between discontinuation of excluded item and study start)
* Clinically significant or unstable cardiovascular, gastrointestinal, hepatic, or renal disease states defined as requiring on-going changes to medication or medical management
* Consumption of smoking or chewing tobacco, or other nicotine-containing products for >1 day per week
* Consumption of >14 alcohol drinks per week
* Pregnant, breastfeeding, or plan to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change between intervention arms in baseline adjusted LDL-c at 4 weeks | 4 weeks
  Change in LDL-c
Change between intervention arms in baseline adjusted TMAO at 4 weeks | 4 weeks
  Change in TMAO

SECONDARY OUTCOMES:
Change between intervention arms in baseline adjusted LDL-c at 8 weeks | 8 weeks
  Change in LDL-c
Change between intervention arms in baseline adjusted LDL-c at 12 weeks | 12 weeks
  Change in LDL-c
Change between intervention arms in baseline adjusted TMAO at 8 weeks | 8 weeks
  Change in TMAO
Change between intervention arms in baseline adjusted TMAO at 12 weeks | 12 weeks
  Change in TMAO
Change between intervention arms in baseline adjusted lipid panel parameters at 4 weeks | 4 weeks
  Change in lipid panel
Change between intervention arms in baseline adjusted lipid panel parameters at 8 weeks | 8 weeks
  Change in lipid panel
Change between intervention arms in baseline adjusted lipid panel parameters at 12 weeks | 12 weeks
  Change in lipid panel
Change between intervention arms in baseline adjusted BMI at 4 weeks | 4 weeks
  Weight and height will be combined to report BMI in kg/m^2
Change between intervention arms in baseline adjusted BMI at 8 weeks | 8 weeks
  Weight and height will be combined to report BMI in kg/m^2
Change between intervention arms in baseline adjusted BMI at 12 weeks | 12 weeks
  Weight and height will be combined to report BMI in kg/m^2
Change between intervention arms in baseline adjusted blood pressure at 4 weeks | 4 weeks
  Measured with Sphygmocor device, both systolic and diastolic blood pressures
Change between intervention arms in baseline adjusted blood pressure at 8 weeks | 8 weeks
  Measured with Sphygmocor device, both systolic and diastolic blood pressures
Change between intervention arms in baseline adjusted blood pressure at 12 weeks | 12 weeks
  Measured with Sphygmocor device, both systolic and diastolic blood pressures
Change between intervention arms in baseline adjusted hemoglobin A1c at 4 weeks | 4 weeks
  Change in hemoglobin A1c
Change between intervention arms in baseline adjusted hemoglobin A1c at 8 weeks | 8 weeks
  Change in hemoglobin A1c
Change between intervention arms in baseline adjusted hemoglobin A1c at 12 weeks | 12 weeks
  Change in hemoglobin A1c

OTHER OUTCOMES:
Difference between intervention arms in baseline adjusted gut microbiome at 4 weeks | 4 weeks
  Change in alpha diversity
Change between intervention arms in baseline adjusted gut microbiome at 8 weeks | 8 weeks
  Change in alpha diversity
Change between intervention arms in baseline adjusted gut microbiome at 12 weeks | 12 weeks
  Change in alpha diversity
Change between intervention arms in baseline adjusted complete blood count | 12 weeks
  Change in complete blood count
Change between intervention arms in baseline adjusted serum C-reactive protein | 12 weeks
  Change in C-reactive protein
Change between intervention arms in baseline adjusted serum high sensitivity C-reactive protein | 12 weeks
  Change in high sensitivity C-reactive protein
Change between intervention arms in baseline adjusted serum vitamin B12 level | 12 weeks
  Change in vitamin B12
Change between intervention arms in baseline adjusted serum iron | 12 weeks
  Change in serum iron
Change in calorie intake | 12 weeks
  Change in calorie intake
Change in meal patterns post vegan meal kit intervention | 12 weeks
  Change in percent of vegan meals per week

CONTACTS AND LOCATIONS:
Locations (1):
- David Grant U.S. Air Force Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Vegan Diet. National Health Service website. Updated Aug 2018. Accessed 10 Jan 2021.
- [Background] Najjar RS, Moore CE, Montgomery BD. A defined, plant-based diet utilized in an outpatient cardiovascular clinic effectively treats hypercholesterolemia and hypertension and reduces medications. Clin Cardiol. 2018 Mar;41(3):307-313. doi: 10.1002/clc.22863. Epub 2018 Mar 25. PMID 29575002
- [Background] Heianza Y, Ma W, Manson JE, Rexrode KM, Qi L. Gut Microbiota Metabolites and Risk of Major Adverse Cardiovascular Disease Events and Death: A Systematic Review and Meta-Analysis of Prospective Studies. J Am Heart Assoc. 2017 Jun 29;6(7):e004947. doi: 10.1161/JAHA.116.004947. PMID 28663251
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Wang Z, Bergeron N, Levison BS, Li XS, Chiu S, Jia X, Koeth RA, Li L, Wu Y, Tang WHW, Krauss RM, Hazen SL. Impact of chronic dietary red meat, white meat, or non-meat protein on trimethylamine N-oxide metabolism and renal excretion in healthy men and women. Eur Heart J. 2019 Feb 14;40(7):583-594. doi: 10.1093/eurheartj/ehy799. PMID 30535398
- [Background] Crimarco A, Springfield S, Petlura C, Streaty T, Cunanan K, Lee J, Fielding-Singh P, Carter MM, Topf MA, Wastyk HC, Sonnenburg ED, Sonnenburg JL, Gardner CD. A randomized crossover trial on the effect of plant-based compared with animal-based meat on trimethylamine-N-oxide and cardiovascular disease risk factors in generally healthy adults: Study With Appetizing Plantfood-Meat Eating Alternative Trial (SWAP-MEAT). Am J Clin Nutr. 2020 Nov 11;112(5):1188-1199. doi: 10.1093/ajcn/nqaa203. PMID 32780794
- [Background] Koeth RA, Wang Z, Levison BS, Buffa JA, Org E, Sheehy BT, Britt EB, Fu X, Wu Y, Li L, Smith JD, DiDonato JA, Chen J, Li H, Wu GD, Lewis JD, Warrier M, Brown JM, Krauss RM, Tang WH, Bushman FD, Lusis AJ, Hazen SL. Intestinal microbiota metabolism of L-carnitine, a nutrient in red meat, promotes atherosclerosis. Nat Med. 2013 May;19(5):576-85. doi: 10.1038/nm.3145. Epub 2013 Apr 7. PMID 23563705